CLINICAL TRIAL: NCT04324372
Title: An Open Label Multicentric Phase 1 Study of HEC68498 in Patients With Advanced Refractory Solid Tumors.
Brief Title: Clinical Study of HEC68498 in Patients With Advanced Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEC68498-P-01
Record Dates: First submitted 2020-03-18; First posted 2020-03-27 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Advanced Refractory Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HEC68498 (Experimental): HEC68498 will be administered daily
  Interventions: Drug: HEC68498

INTERVENTIONS:
Drug: HEC68498 — HEC68498 is a potent,highly selective inhibitor of class 1 isozymes of phosphoinositide 3-kinase/mammalian(PI3K) and of the mammalian target of rapamycin (mTOR). It has shown good activity against fibrosis and inflammation in vitro and in vivo, with a lower effective dose and better efficacy than pirfenidone and nintedanib.

SUMMARY:
Clinical study of HEC68498 in patients with advanced refractory solid tumors. The primary objective is to determine the maximum tolerated dose and dose limiting toxicity of HEC68498 in patients with advanced refractory solid tumors

DETAILED DESCRIPTION:
An open label multicentric Phase 1 study of HEC68498 in patients with advanced refractory solid tumors.The study will follow a 3+3 design until significant toxicity as described in the protocol and considering pharmacokinetics of the study drug determined from cohorts.

ELIGIBILITY:
Inclusion Criteria:

（1）Target subjects

1. 18 years of age ≤ age ≤ 70 years of age, regardless of gender;
2. Patients with various types of advanced solid tumors confirmed by cytological or histological examination.

   Dose escalation test phase: including breast cancer, colorectal cancer, neuroendocrine tumors, etc .; Extended trial phase: limited to patients with HR + / HER2-, triple-negative, breast, colorectal, and neuroendocrine tumors, and patients with HR + / HER2- and colorectal cancer need genetic testing (blood and / or tumor tissue) PIK3CA mutations have been confirmed. Patients with triple negative breast cancer need genetic testing (blood and / or tumor tissue) to confirm PIK3CA / PTEN- mutations.
3. Requires at least standard treatment failure or no standard treatment. Definition of treatment failure: a. Disease progression during or after treatment must have clear imaging or clinical evidence; b. Withdrawal from treatment due to intolerable response.
4. According to the solid tumor evaluation criteria (RECIST 1.1), there is at least one measurable lesion.
5. Relieve from previous chemotherapy, hormone therapy, targeted therapy, radiotherapy or surgical treatment of toxic reactions (according to CTCAE v5.0 grading ≤ 1 except hair loss)
6. ECOG score is 0 or 1 (see Annex 2 for ECOG score criteria);
7. Expected survival time ≥ 12 weeks;

(2) The subject must have proper organ function

1. Blood routine: absolute neutrophil (ANC) ≥ 1.5 × 109 / L; platelet (PLT) ≥ 75 × 109 / L; hemoglobin (Hb) ≥ 90 g / L; Have received hematopoietic cell colony-stimulating growth factors (eg G-CSF, GM-CSF) or have not received blood transfusions. Erythropoietin or erythropoietin therapy can be maintained if it is used immediately before enrollment.
2. Liver function: ALT and AST ≤ 2.5 × ULN (for patients with liver metastases, ALT and AST can be relaxed to ≤ 5.0 × ULN); serum bilirubin ≤ 1.5 × ULN;
3. Renal function: serum creatinine ≤ 1.5 × ULN; or creatinine clearance (CrCl) ≥ 60 mL / min calculated according to the Cockcroft-Gault formula:

   Urine routine urinary protein ≤ 1+; if urinary routine urinary protein ≥ 2+, a 24-hour urine protein quantification is less than 1 g.
4. Electrolyte: LLN ≤ blood potassium ≤ ULN;
5. Coagulation function: international standardized ratio (INR) ≤ 1.5 × ULN; activated partial thromboplastin time (APTT) ≤ 1.5 × ULN; prothrombin time (PT) ≤ 1.5 × ULN;

Exclusion Criteria:

(1) previous treatment history

1. Have previously been treated with PI3K inhibitors, mTOR inhibitors (such as everolimus) or AKT inhibitors.
2. Patients who have received targeted therapy within 4 weeks before the first dose or ≤ 5 × drug half-life (if the half-life of the drug is specified, it is calculated as 5 times the half-life, otherwise 4 weeks);
3. Patients who have received chemotherapy, hormonal antitumor therapy, immunotherapy or major surgery within 4 weeks before the first dose.

   Note: If the previous treatment was nitrosourea or mitomycin, the treatment must be discontinued at least 6 weeks before the first study drug is administered.
4. Patients who have received radiation therapy within 4 weeks before the first dose.
5. Have received clinical trial drug treatment within 4 weeks before the first medication, or are receiving other clinical trial drug treatment;

(2) History of disease and surgery

1. CNS metastases requiring current treatment or uncontrolled CNS metastases; or CNS metastases confirmed but not stable for more than 4 weeks after treatment;
2. Patients with spinal cord compression, cancerous meningitis, or meningitis;
3. Currently diagnosed with type I or type II diabetes or fasting blood glucose levels> 6.7 mmol / L, or HbA1c> 7%;
4. Patients with hypertension controlled by two or more drugs, or uncontrolled hypertension (systolic blood pressure> 140 mmHg or diastolic blood pressure> 90 mmHg);
5. Left ventricular ejection fraction (LVEF) <50%; QTcF> 450 ms for men, QTcF> 470 ms for women (QTcF is calculated using Fridericia's correction formula QTcF = QT / RR 0.33); any room with obvious clinical significance History of arrhythmia (such as ventricular tachycardia, ventricular fibrillation, torsional ventricular tachycardia or frequent ventricular premature beats, congenital prolonged QT interval syndrome).
6. Multiple factors affecting oral medication (eg, inability to swallow, chronic diarrhea, and intestinal obstruction, etc.);
7. Patients with a clear tendency to gastrointestinal bleeding, including the following: local active ulcer lesions and positive fecal occult blood; those with a history of melena and vomiting within 2 months before the first medication; researchers believe that digestion may occur Major bleeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-03-26 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | 28 days
  Patients will receive study drug on a daily basis for 28 days according to the dose and schedule specified for a particular cohort of therapy. Toxicities observed in Cycle 0&1 will be considered for dose limiting toxicity (DLT) and Maximum tolerated dose (MTD)determination

SECONDARY OUTCOMES:
Number of subject with adverse events | up to 4 weeks after last dose
  The toxic effects of the drug would be assessed from adverse events, vital signs and by clinically significant changes in the laboratory evaluations.
Objective response | up to approximately 24 months
  Evaluation of Response: Clinical responses will be presented patient wise for different dose levels.
AUC0-∞ | up to approximately 4 weeks
  area under the concentration versus time curve (AUC) from time zero to infinity
AUC0-t | up to approximately 4 weeks
  AUC from time zero to the time of the last quantifiable concentration time zero to the time of the last quantifiable concentration
Cmax | up to approximately 4 weeks
  maximum observed plasma concentration
tmax | up to approximately 4 weeks
  time of the maximum observed plasma concentration
t½ | up to approximately 4 weeks
  apparent terminal elimination half-life
Vz/F | up to approximately 4 weeks
  apparent volume of distribution

CONTACTS AND LOCATIONS:
Locations (1):
- The Fifth Medical Center of PLA Ceneral Hospital, Beijing, China/BEIJING, China

IPD SHARING:
Plan to Share IPD: No